CLINICAL TRIAL: NCT04263454
Title: The Innate Central Nervous System Immune Response to an Experimental Immune Challenge in People With Fibromyalgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Fibromyalgia Syndrome Association (Other)
Responsible Party: Principal Investigator, Jarred Younger, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB-140930002
Record Dates: First submitted 2020-02-03; First posted 2020-02-10 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Fibromyalgia
Keywords: neuroinflammation; neuroimaging; fibromyalgia; endotoxin; chronic pain
MeSH Terms: conditions — Fibromyalgia; Neuroinflammatory Diseases; Chronic Pain | interventions — endotoxin, Escherichia coli; Endotoxins; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Healthy controls and fibromyalgia patients will have an MRI scan both before and 3 hours post endotoxin injection.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Control (Other): All healthy control participants will undergo the same screening and experimental procedures. Healthy controls must report no other medical conditions ( including fibromyalgia) to be considered for inclusion. All healthy controls will have an MRI scan performed both before and 3 hours post 0.4ng/kg endotoxin injection.
  Interventions: Drug: Endotoxin, Escherichia Coli; Procedure: Magnetic Resonance Spectroscopy
- Fibromyalgia (Experimental): All fibromyalgia participants will undergo the same screening and experimental procedures. However, fibromyalgia participants will need to meet 2010 American College of Rheumatology diagnostic criteria for fibromyalgia. All fibromyalgia participants will have an MRI scan performed both before and 3 hours post 0.4ng/kg endotoxin injection.
  Interventions: Drug: Endotoxin, Escherichia Coli; Procedure: Magnetic Resonance Spectroscopy

INTERVENTIONS:
Drug: Endotoxin, Escherichia Coli — Endotoxin is a purified lipopolysaccharide prepared from E. coli O:113 and vialed under good manufacturing practice guidelines.
  Other Names: Endotoxin
Procedure: Magnetic Resonance Spectroscopy — MRI is a non-invasive imaging technique and does not utilize ionizing radiation.
  Other Names: MRI

SUMMARY:
The major goal of this study is to determine if the innate immune response is dysregulated in people with fibromyalgia, compared to healthy controls. Magnetic resonance spectroscopy will be used to measure changes in the brain's metabolic profile following an experimental immune stimulus, to test whether individuals with fibromyalgia show a heightened immune response in the brain. The ultimate goal of this research is to better understand the role of brain inflammation in the pathophysiology of chronic pain and fatigue, which will guide the development of more effective therapies for these conditions.

DETAILED DESCRIPTION:
The study consists of two sessions: the screening session and the experimental session. During the initial phone screening, individuals who contact the study team will be given information about the study, including a description of all study-related procedures. If interested, participants will then be taken through a phone screen interview that will ask them to report demographic information (date of birth, race, ethnicity), height and weight, and list of medical conditions and current medications, surgical history within the past year, amount of weekly consumption of alcohol, tobacco products, and illicit substances, viral or bacterial infections within the past 3 months, recent vaccines received, and current participation in other research. The standard MRI Safety form will be administered to ensure participants do not have ferromagnetic implants or other contraindications to MRI (e.g. claustrophobia).A self-report will also be administered to ascertain that potential fibromyalgia participants meet 2016 American College of Rheumatology (ACR) criteria for fibromyalgia. The phone screen is intended to reduce participant burden by identifying exclusion criteria without the need to attend at UAB. Participants who meet initial screening criteria will be invited to attend an in-person screening visit.

During the screening visit, participants will go to the Clinical Research Unit (CRU) on the 15th floor of Jefferson Tower. Participants will be asked to fast prior to this visit. Participants will provide written informed consent before any study procedures are initiated. Participants will provide a urine sample for pregnancy testing. Vital signs (blood pressure, heart rate), aural temperature, height and weight will be measured and recorded. Participants will undergo 12-lead electrocardiogram and provide a maximum of 60cc of blood into labeled blood collection tubes for screening tests. A tender point exam will be administered to assess fibromyalgia symptomatology. The procedure uses a pressure algometer, a hand-held instrument with a small rubber tip that is applied to the participant's skin over standardized regions of the body (occipital, low cervical, upper trapezius, supraspinatus, anterior second rib, lateral epicondyle, gluteal, greater trochanteric, or medial knee). Pressure is slowly increased at a constant rate until the participant reports the sensation changing from one of pressure to one of pain or discomfort. Participants will complete a demographics form , Brief Pain Inventory, Fibromyalgia Impact Questionnaire, Multidimensional Fatigue Inventory, and Multiple Abilities Symptom Questionnaire. The blood will be tested by the UAB Hospital Labs to ensure that the participant meets the study criteria. The ECG will be forwarded to the study physician who will assess for evidence of conduction abnormalities or of ischemia. If the blood tests or ECG are abnormal, the study physician will determine if the participant should be advised to see their PCP. Following availability of all results from the screening visit, participants will be contacted via phone and informed of their eligibility to attend the experimental session.

During the experimental session, the administration of endotoxin, brain imaging, and related procedures will be performed at the CRU. No fasting is required prior to this visit, and participants will be asked to eat breakfast prior to arrival and will be provided with meal suggestions. Baseline vital sign measurements consisting of resting blood pressure and pulse rate will be measured and recorded within 60 minutes prior to the start of imaging. ECG and pregnancy tests will be repeated and participants will be excluded from participation in the session if conduction abnormalities are found (same criteria as used during screening) or if participants are found to be pregnant. Participants will undergo MRI imaging for approximately 1 hour. Participants will leave the scanner and complete questionnaire measures assessing participant's current level of fatigue, pain, and mood symptoms. Grip strength will also be assessed. A low dose of endotoxin (0.3ng/kg) will then be administered by the study nurse via intravenous infusion. Vital signs will be periodically monitored for the rest of the session. Participants will remain in the laboratory for three hours before being placed into the MRI scanner to complete a second, identical, imaging session. The self-report questionnaire measures and grip strength will be repeated every hour following endotoxin administration in order to quantify changes in symptoms due to LPS. To avoid participant discomfort and to optimize study integrity, a standardized meal of approximately 600-kcal will be provided to each participant between the two MRI sessions, as well as a later snack of approximately 200-kcal. The meal is standardized to caloric quantity and timing to offset any effects of food intake on the immune response.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Age 18-55, inclusive;
* Adequate English for study participation;
* (fibromyalgia group only) Meet 2010 American College of Rheumatology criteria for the diagnosis of fibromyalgia
* Able to undergo IV cannulation and to provide the requisite blood samples;
* BMI 18-39.9 inclusive;
* Resting heart rate ≥55
* Supine systolic blood pressure of <140mmHg and >100mmHg AND
* Diastolic blood pressure <90mgHG and >60mmHg at screening.

Exclusion Criteria:

* Cardiovascular, immune or infectious disease (e.g. HIV, HCV), or diabetes;
* At screening, a 12-lead ECG demonstrating QTc>450 or QRS >120msec. If the QTc exceeds 450msec, or QRS exceeds 120msec, the ECG will be repeated x2 and the median of the three values will be used to determine the participant's eligibility.
* Rheumatologic or autoimmune disease;
* Vaccine administered within 4 weeks of study participation;
* Viral or bacterial illness requiring medical attention and/or antibiotics within 3 months of study participation, or any illness or fever within 1 month of study participation;
* Surgical procedure within 3 months of study participation;
* Regular use of anti-inflammatory of immunomodulatory drugs (occasional use of NSAIDs is not an exclusion as long as the participant does not administer within 5 days of study participation);
* Current use of opioid medication;
* Current smoker or ceased smoking ≤12 months prior to participation;
* High alcohol consumption;
* Consumption of drugs of abuse (except alcohol);
* Significant psychological comorbidity that in the discretion of the investigator compromises study integrity;
* Current participation in any other research;
* Ongoing litigation or worker's compensation claim;
* Hospital Anxiety and Depression score indicating clinically significant depression;
* Currently pregnant or positive screening urine pregnancy test;
* Complete blood count values outside the normal clinical ranges, erythrocyte sedimentation rate (ESR) >60, C-reactive protein (CRP) >3, positive rheumatoid factor (RHF), or positive antinuclear antibodies (ANA).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jarred M Younger, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Control: Healthy controls must report no other medical conditions (including fibromyalgia) to be considered for inclusion. All healthy controls will have an MRI scan performed both before and 3 hours post 0.4ng/kg endotoxin injection.
  Endotoxin, Escherichia Coli: Endotoxin is a purified lipopolysaccharide prepared from E. coli O:113 and vialed under good manufacturing practice guidelines.
  Magnetic Resonance Spectroscopy: MRI is a non-invasive imaging technique and does not utilize ionizing radiation.
- Fibromyalgia: Fibromyalgia participants will need to meet 2010 American College of Rheumatology diagnostic criteria for fibromyalgia. All fibromyalgia participants will have an MRI scan performed both before and 3 hours post 0.4ng/kg endotoxin injection.
  Endotoxin, Escherichia Coli: Endotoxin is a purified lipopolysaccharide prepared from E. coli O:113 and vialed under good manufacturing practice guidelines.
  Magnetic Resonance Spectroscopy: MRI is a non-invasive imaging technique and does not utilize ionizing radiation.
Period: Overall Study
Arm/Group | Healthy Control | Fibromyalgia
Started | 16 | 20
Completed | 13 | 12
Not Completed | 3 | 8
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 3 | 5
Not completed — Poor Data Quality | 0 | 1

BASELINE CHARACTERISTICS:
Population: analysis population as defined in participant flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Fibromyalgia | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (10.5) | 42.6 (10.2) | 41.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 7 | 10 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
Pain Severity [Mean (Standard Deviation); unit: units on a scale] — 0 to 10 scale (higher is worse)
  units on a scale | 0.15 (0.38) | 6.25 (0.45) | 3.2 (.41)
Fatigue Severity [Mean (Standard Deviation); unit: units on a scale] — 0 to 10 scale (higher is worse)
  units on a scale | 1.00 (1.23) | 7.17 (1.59) | 4.09 (1.41)

OUTCOME MEASURES:

1. Primary Outcome: Change in Ratio of Choline/ Creatine (CHO/CR) in the Brain From Baseline to 3 Hrs Post-endotoxin Administration
Description: The concentration of brain metabolite CHO will be measured via MRI scan as a measure of neuroinflammation. This measurement will be performed in both the control and experimental group. Increased CHO is a marker of increased cell turnover that can be seen during neuroinflammation.
Time Frame: 3 hours (From Baseline to 3 Hrs Post-endotoxin Administration)
Population: as defined in participant flow
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Healthy Control | Fibromyalgia
Number analyzed (Participants) | 13 | 12
ratio | -.0021 (.01664) | -.0058 (.01465)

2. Primary Outcome: Change in Ratio of Myoinositol/ Creatine (MI/CR) in the Brain From Baseline to 3hrs Post-endotoxin Administration
Description: The concentration of brain metabolite MI will be assessed via MRI scan as a measure of neuroinflammation. This measurement will be performed in both the control and experimental group. MI is a marker of microglia, and an acute increase in this metabolite could indicate microglia proliferation or accumulation.
Time Frame: 3 hours (From Baseline to 3 Hrs Post-endotoxin Administration)
Population: as defined in participant flow
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Healthy Control | Fibromyalgia
Number analyzed (Participants) | 13 | 12
ratio | -.0049 (.31164) | .1030 (.18022)

3. Primary Outcome: Change in Brain Temperature From Baseline to 3 Hours Post-endotoxin Administration.
Description: The temperature of the brain will be assessed via MRI scan as a measure of neuroinflammation. This measurement will be performed in both the control and experimental group. Increased brain temperature certain areas may indicate an abnormally increased inflammatory response.
Time Frame: 3 hours (From Baseline to 3 Hrs Post-endotoxin Administration)
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Healthy Control | Fibromyalgia
Number analyzed (Participants) | 13 | 12
degrees Celsius | 0.10 (0.44) | 0.55 (0.55)

ADVERSE EVENTS:
Time Frame: Participants were observed in the research setting for 10 hours.
Description: CT.gov definitions are used for adverse events.
Arm/Group | Healthy Control | Fibromyalgia
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT04263454/Prot_002.pdf
  • Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT04263454/SAP_003.pdf